CLINICAL TRIAL: NCT03266146
Title: The Efficacy and Safety of 36 Weeks Short-Term Optimization Treatment of Glucocorticosteroid in the Patients With Chronic Recurrent Drug-Induced Liver Injury
Brief Title: 36 Weeks Short-Term Optimization Treatment of Glucocorticosteroid in the Patients With Chronic Recurrent DILI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJ302-FGRXGB-003
Record Dates: First submitted 2017-08-26; First posted 2017-08-29 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Drug-induced Liver Injury,Chronic
Keywords: Drug-induced Liver Injury; Recurrence; Methylprednisolone; Short-term
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury, Chronic; Chemical and Drug Induced Liver Injury; Recurrence | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 36 Weeks Methylprednisolone (Experimental): Participants in 36 weeks of glucocorticoid treatment group will receive methylprednisolone, 48mg/d for the 1st week, 32mg/d for the 2nd week, 24mg/d for the next two weeks, followed by 16mg/d for 20 weeks and reduction in doses of methylprednisolone by 4 mg per 4 weeks until drug withdrawal. Participants in 36 weeks of glucocorticoid treatment group also will receive standard treatment including reduced glutathione, glycyrrhizin, ademetionine, alprostadil, or ursodeoxycholic acid (UDCA). Participants will then be followed for 24 weeks.
  Interventions: Drug: 36 Weeks Methylprednisolone
- 48 Weeks Methylprednisolone (Experimental): Participants in 48 weeks of glucocorticoid treatment group will receive methylprednisolone, 48mg/d for the 1st week, 32mg/d for the 2nd week, 24mg/d for the next two weeks, followed by 16mg/d for 32 weeks and reduction in doses of methylprednisolone by 4 mg per 4 weeks until drug withdrawal. Participants in glucocorticoid 48 weeks of treatment group also will receive standard treatment including reduced glutathione, glycyrrhizin, ademetionine, alprostadil, or ursodeoxycholic acid (UDCA). Participants will then be followed for 24 weeks.
  Interventions: Drug: 48 weeks Methylprednisolone

INTERVENTIONS:
Drug: 36 Weeks Methylprednisolone — Participants in 36 weeks of glucocorticoid treatment group will receive methylprednisolone, 48mg/d for the 1st week, 32mg/d for the 2nd week, 24mg/d for the next two weeks, followed by 16mg/d for 20 weeks and reduction in doses of methylprednisolone by 4 mg per 4 weeks until drug withdrawal. Participants in 36 weeks of glucocorticoid treatment group also will receive standard treatment including reduced glutathione, glycyrrhizin, ademetionine, alprostadil, or ursodeoxycholic acid (UDCA).The total treatment duration will be 36 weeks. Follow-up duration is 24 weeks.
  Other Names: MEDROL,NDC0009-0056-02
  Arms: 36 Weeks Methylprednisolone
Drug: 48 weeks Methylprednisolone — Participants in 48 weeks of glucocorticoid treatment group will receive methylprednisolone, 48mg/d for the 1st week, 32mg/d for the 2nd week, 24mg/d for the next two weeks, followed by 16mg/d for 32 weeks and reduction in doses of methylprednisolone by 4 mg per 4 weeks until drug withdrawal. Participants in 36 weeks of glucocorticoid treatment group also will receive standard treatment including reduced glutathione, glycyrrhizin, ademetionine, alprostadil, or ursodeoxycholic acid (UDCA).The total treatment duration will be 48 weeks. Follow-up duration is 24 weeks.
  Other Names: MEDROL,NDC0009-0056-02
  Arms: 48 Weeks Methylprednisolone

SUMMARY:
This study is to observe the efficacy and safety of 36 weeks short-term optimization treatment of glucocorticosteroid in the patients with chronic recurrent drug-induced liver injury (DILI).

DETAILED DESCRIPTION:
Drug-induced liver injury (DILI) refers to liver diseases caused by drugs and toxic substances. DILI is a clinical event that can be associated with severe outcomes such as acute liver failure. Up to now, approximately 1100 drugs, herbal products, vitamins and illicit compounds are associated with liver injury. Recently, the incidence of DILI is rising. In our hospital, hospitalized patients with DILI was increased from 1.39% in 2002 to 2.31% in 2006, and further up to 3.17% in 2011, which indicated 2.3-folds increase over last ten years. About 20% patients with acute DILI are prone to chronic liver disease. For patients with chronic recurrent DILI, routine liver protective treatment was difficult to rescue abnormal liver functions. Moreover, increasing health care costs seriously affect the patient's quality of life. Glucocorticosteroids can inhibit the non-specific inflammation and permeability of the capillary bile duct, limit the activation of T lymphocytes, and selectively inhibit B lymphocytes to produce antibodies, thus preventing or delaying the immune-induced liver injury. In our pre-clinical trials (NCT02651350), we found that the rate of recurrence of the glucocorticoid treatment group was significant lower (<10%) than the control group (about 50%) (P <0.001) and there was significant difference of liver histological change during baseline and treatment end between the glucocorticoid treatment group and the control group. Meanwhile, we did not find obvious glucocorticoid's side effect in the glucocorticoid treatment group. At the same time, we found that there was good effect in 36 weeks glucocorticoid treatment in several patients. Therefore, we shall design two groups on the basis of the ratio of 1:1, namely, 36 weeks of glucocorticoid treatment group and 48 weeks of glucocorticoid treatment group in order to evaluate the efficacy and safety of 36 weeks short-term optimization treatment of glucocorticosteroid in the patients with chronic recurrent DILI.

Participants in 36 weeks of glucocorticoid treatment group will receive methylprednisolone, 48mg/d for the 1st week, 32mg/d for the 2nd week, 24mg/d for the next two weeks, followed by 16mg/d for 20 weeks and reduction in doses of methylprednisolone by 4 mg per 4 weeks until drug withdrawal. Participants in 36 weeks of glucocorticoid treatment group also will receive standard treatment including reduced glutathione, glycyrrhizin, ademetionine, alprostadil, or ursodeoxycholic acid (UDCA).Participants will then be followed for 24 weeks. Participants in 48 weeks of glucocorticoid treatment group will receive methylprednisolone, 48mg/d for the 1st week, 32mg/d for the 2nd week, 24mg/d for the next two weeks, followed by 16mg/d for 32 weeks and reduction in doses of methylprednisolone by 4 mg per 4 weeks until drug withdrawal. Participants in glucocorticoid 48 weeks of treatment group also will receive standard treatment including reduced glutathione, glycyrrhizin, ademetionine, alprostadil,or ursodeoxycholic acid (UDCA).Participants will then be followed for 24 weeks.

The efficacy and safety of 36 weeks short-term optimization treatment of glucocorticosteroid in the patients with chronic recurrent DILI will be observed and compared with 48 weeks glucocorticosteroid treatment during the treatment and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Meet with ACG clinic guidelines for diagnostic criteria of chronic DILI;
2. The time of recurrence is 1 or more than 1;

   The definition of recurrence, meet any of the following conditions:
   * the level of serum AST or ALT is elevated more than 5 fold ULN;
   * the level of serum AST or ALT is two times higher than before;
3. Meet any of the following conditions:

   * serum AST or ALT ≥ 10 fold ULN;
   * serum AST or ALT ≥ 5 fold ULN and TBIL ≥ 2 fold ULN;
   * liver histology indicates bridging necrosis or multiacinar necrosis or moderate or more inflammation or inflammation G3 or more;
4. Women of childbearing age had a negative urine pregnancy test, and the subjects are willing to have no family planning during the study and to take effective measures;
5. Voluntary participation, understanding and signing of informed consent, comply with the requirements of the research.

   -

Exclusion Criteria:

1. Patients with serious pre-existent comorbid conditions (vertebral compression fractures,psychosis,active peptic ulcer, brittle diabetes,uncontrolled hypertension;
2. Patients with intolerances to prednisone;
3. Patients with severe infection receiving antibiotics, anti-fungal,anti-viral therapy;
4. Viral hepatitis,alcoholic or non-alcoholic liver disease,Wilson's disease or other inherited metabolic liver diseases.
5. Pregnancy or desire of pregnancy;
6. Breast-feeding;
7. Liver cancer or other malignant tumor.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2017-09-02 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Recurrence rate of illness, namely, appearance of obviously abnormal liver function again during treatment and follow-up period. The definition of recurrence: The level of AST or ALT is elevated more than 5 fold ULN or is two times higher than before. | From week 1 to week 60 or 72
  To analyze the clinical efficacy of glucocorticosteroid treatment

SECONDARY OUTCOMES:
The liver histological changes between two liver biopsies (baseline and treatment end) | At week 0 and at week 36 week or 48 week
  To analyze the clinical efficacy of glucocorticosteroid treatment
Days of normalization or falling by half compared to admission of liver functions including serum levels of ALT, AST, TBIL,GGT and ALP. | From week 1 to week 36 or 48
  To analyze the clinical efficacy of glucocorticosteroid treatment

CONTACTS AND LOCATIONS:
Overall Officials: Zhengsheng Zou, Dr., Principal Investigator — Beijing 302 Hospital,China.
Locations (1):
- Beijing 302 hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chalasani NP, Hayashi PH, Bonkovsky HL, Navarro VJ, Lee WM, Fontana RJ; Practice Parameters Committee of the American College of Gastroenterology. ACG Clinical Guideline: the diagnosis and management of idiosyncratic drug-induced liver injury. Am J Gastroenterol. 2014 Jul;109(7):950-66; quiz 967. doi: 10.1038/ajg.2014.131. Epub 2014 Jun 17. PMID 24935270
- [Background] Moreno L, Sanchez-Delgado J, Vergara M, Casas M, Miquel M, Dalmau B. Recurrent drug-induced liver injury (DILI) with ciprofloxacin and amoxicillin/clavulanic. Rev Esp Enferm Dig. 2015 Dec;107(12):767-8. doi: 10.17235/reed.2015.3810/2015. PMID 26671593
- [Background] Tencate V, Komorowski R, Cronin D, Hong J, Gawrieh S. A case study: refractory recurrent autoimmune hepatitis following liver transplantation in two male patients. Transplant Proc. 2014 Jan-Feb;46(1):298-300. doi: 10.1016/j.transproceed.2013.09.028. PMID 24507072
- [Background] Lucena MI, Kaplowitz N, Hallal H, Castiella A, Garcia-Bengoechea M, Otazua P, Berenguer M, Fernandez MC, Planas R, Andrade RJ. Recurrent drug-induced liver injury (DILI) with different drugs in the Spanish Registry: the dilemma of the relationship to autoimmune hepatitis. J Hepatol. 2011 Oct;55(4):820-7. doi: 10.1016/j.jhep.2010.12.041. Epub 2011 Feb 19. PMID 21338638
- [Background] Suzuki A, Brunt EM, Kleiner DE, Miquel R, Smyrk TC, Andrade RJ, Lucena MI, Castiella A, Lindor K, Bjornsson E. The use of liver biopsy evaluation in discrimination of idiopathic autoimmune hepatitis versus drug-induced liver injury. Hepatology. 2011 Sep 2;54(3):931-9. doi: 10.1002/hep.24481. Epub 2011 Aug 8. PMID 21674554
- [Background] Weiler-Normann C, Schramm C. Drug induced liver injury and its relationship to autoimmune hepatitis. J Hepatol. 2011 Oct;55(4):747-9. doi: 10.1016/j.jhep.2011.02.024. Epub 2011 Mar 9. No abstract available. PMID 21396413
- [Background] Bessone F, Lucena MI, Roma MG, Stephens C, Medina-Caliz I, Frider B, Tsariktsian G, Hernandez N, Bruguera M, Gualano G, Fassio E, Montero J, Reggiardo MV, Ferretti S, Colombato L, Tanno F, Ferrer J, Zeno L, Tanno H, Andrade RJ. Cyproterone acetate induces a wide spectrum of acute liver damage including corticosteroid-responsive hepatitis: report of 22 cases. Liver Int. 2016 Feb;36(2):302-10. doi: 10.1111/liv.12899. Epub 2015 Jul 16. PMID 26104271
- [Background] Sugimoto K, Ito T, Yamamoto N, Shiraki K. Seven cases of autoimmune hepatitis that developed after drug-induced liver injury. Hepatology. 2011 Nov;54(5):1892-3. doi: 10.1002/hep.24513. Epub 2011 Aug 9. No abstract available. PMID 21725992
- [Background] Fujiwara K, Yokosuka O. Histological discrimination between autoimmune hepatitis and drug-induced liver injury. Hepatology. 2012 Feb;55(2):657. doi: 10.1002/hep.24768. No abstract available. PMID 22038865
- [Background] Manns MP, Czaja AJ, Gorham JD, Krawitt EL, Mieli-Vergani G, Vergani D, Vierling JM; American Association for the Study of Liver Diseases. Diagnosis and management of autoimmune hepatitis. Hepatology. 2010 Jun;51(6):2193-213. doi: 10.1002/hep.23584. No abstract available. PMID 20513004
- [Background] Fontana RJ, Hayashi PH, Gu J, Reddy KR, Barnhart H, Watkins PB, Serrano J, Lee WM, Chalasani N, Stolz A, Davern T, Talwakar JA; DILIN Network. Idiosyncratic drug-induced liver injury is associated with substantial morbidity and mortality within 6 months from onset. Gastroenterology. 2014 Jul;147(1):96-108.e4. doi: 10.1053/j.gastro.2014.03.045. Epub 2014 Mar 27. PMID 24681128
- [Background] Stine JG, Chalasani NP. Drug Hepatotoxicity: Environmental Factors. Clin Liver Dis. 2017 Feb;21(1):103-113. doi: 10.1016/j.cld.2016.08.008. Epub 2016 Oct 13. PMID 27842766
- [Background] Hayashi PH, Rockey DC, Fontana RJ, Tillmann HL, Kaplowitz N, Barnhart HX, Gu J, Chalasani NP, Reddy KR, Sherker AH, Hoofnagle JH; Drug-Induced Liver Injury Network (DILIN) Investigators. Death and liver transplantation within 2 years of onset of drug-induced liver injury. Hepatology. 2017 Oct;66(4):1275-1285. doi: 10.1002/hep.29283. Epub 2017 Aug 26. PMID 28543844
- [Background] Chalasani N, Bonkovsky HL, Fontana R, Lee W, Stolz A, Talwalkar J, Reddy KR, Watkins PB, Navarro V, Barnhart H, Gu J, Serrano J; United States Drug Induced Liver Injury Network. Features and Outcomes of 899 Patients With Drug-Induced Liver Injury: The DILIN Prospective Study. Gastroenterology. 2015 Jun;148(7):1340-52.e7. doi: 10.1053/j.gastro.2015.03.006. Epub 2015 Mar 6. PMID 25754159
- [Derived] Huang A, Zhu Y, Liu S, Sun Y, Liu Z, Liang QS, Zhao J, Chang BX, Bi JF, Liu JT, Zhai XR, Xie H, Li N, Tian H, Han L, Zhuang Y, Ma H, Teng GJ, Zhang W, Aithal GP, Ji D, Zhao J, Zou Z. An optimized short-term steroid therapy for chronic drug-induced liver injury: A prospective randomized clinical trial. Liver Int. 2024 Jun;44(6):1435-1447. doi: 10.1111/liv.15899. Epub 2024 Mar 14. PMID 38483145